CLINICAL TRIAL: NCT03674996
Title: Safety and Security Evaluation of Patients Submitted to Minimally Invasive Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Discharge after prostatectomy
Record Dates: First submitted 2018-07-21; First posted 2018-09-18 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
Keywords: Prostatectomy; Patient satisfaction; Questionnaire
MeSH Terms: conditions — Prostatic Neoplasms; Patient Satisfaction | interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Same day discharge (Experimental): Patients submitted to minimally invasive radical prostatectomy, and discharged 12 hours after the surgery.
  Interventions: Other: Same day discharge
- Next-day discharge (Experimental): Patients submitted to minimally invasive radical prostatectomy, and discharged 24 hours after the surgery.
  Interventions: Other: Next-day discharge
- 2-days discharge (Other): Patients submitted to minimally invasive radical prostatectomy, and discharged 48 hours after the surgery.
  Interventions: Other: 2-days discharge

INTERVENTIONS:
Other: Same day discharge — Discharge of the patient 12 hours after the minimally invasive radical prostatectomy - experimental group
  Arms: Same day discharge
Other: Next-day discharge — Discharge of the patient 24 hours after the minimally invasive radical prostatectomy - experimental group
  Arms: Next-day discharge
Other: 2-days discharge — Discharge of the patient 24 hours after the minimally invasive radical prostatectomy - control group
  Arms: 2-days discharge

SUMMARY:
This project aims to evaluate safety and security of patients submitted to minimally invasive radical prostatectomy, who received discharge from hospital in the same day of the surgery (Group I), on the 1st post-surgery day (Group II) and in the 2nd post-surgery day (Group III - control). The specific aims are the evaluation of fail index and factors that influence the permanence in the hospital, the satisfaction of patients, the perception of security of patient, the index of post-discharge complications and the costs related to different times of hospitalization. On randomization, those patients in Group I must match the early hospital discharge criteria defined in the study. Thus, they will be forwarded to "Casa de Apoio Madre Paulina", where will receive nursing care until the next day when, in the morning, will be reevaluated in the ambulatory of urology from Barretos Cancer Hospital. The patients of Group II will be evaluated in the ambulatory in the 2nd post-surgery day, before the discharge. In the Group III (control), the patients will be discharged in the 2nd post-surgery day (routine of Barretos Cancer Hospital). All patients who accept to be enrolled in the study will sign the Consent Term previously the surgery. At the 10th post-surgery day, in the follow-up, it will be applied the Patients' Satisfaction with Mental Health Services Scale (SATIS-BR) questionnaire and an inventory. The data will be descriptive considering average, standard deviation, minimum and maximum value and quartile to the quantitative variables and frequency tables to the qualitative variables. In order to determine the groups' homogeneity, some sociodemographic and clinical characteristics will be compared. To the qualitative variables, it will be used chi-squared test (of Fishers exact test), and to the quantitative variables it will be used variance analysis (or Kruskal-Wallis test). The patients' satisfaction will be measured using SATIS-BR, which consists in three numeric domains (ranging from 1 to 5). The comparison of each domain among the groups will be performed using ANOVA. Then, linear regression will be performed in order to analyze the relationship of the patients' characteristics influencing the satisfaction. The rates of fail, clinical security, security perception and post-discharge complications will be compared among the groups using chi-squared test (of Fisher's exact test). There will be considered the significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Localized Prostate Cancer
* BMI ≤ 35
* Specific Prostate Antigen ≤ 30 ng/ml
* Gleason score ≤ 7
* Hemoglobin ≤ 12g/dl
* American Society of Anesthesiologists Score ≤ 2
* Absence of psychiatric disease

Exclusion Criteria:

* Perioperative results with estimated blood loss > 750 ml
* Blood transfusion need
* Operative time > 4 hours
* Nausea or vomiting at the discharge
* Uncontrollable pain at the discharge
* Postural hypotension

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Satisfaction of the patients: SATIS-BR | 48 months
  This outcome will be evaluated through SATIS-BR questionnaire
  The unabbreviated scale name is "Escala da avaliação da satisfação dos usuários " ("Scale of evaluation of satisfaction of patients", in free English). The questionnaire contains 39 questions, with possible answers arranged in a Likert scale of 5 points, in which the value 1 indicates the lowest degree of satisfaction (worst outcome) and the value 5 indicates the highest degree of satisfaction (best outcome) with the service. The analysis will be performed in each question individually. The comparison of each question among groups will be performed using Analysis of Variance (ANOVA). Subsequently, Linear Regression will be used to verify the joint relationship among the characteristics of patients with the group influencing satisfaction.
  Additionally, there are 5 qualitative questions that will be analyzed in relation to factors that influence hospital stay and factors that influence the patients' satisfaction.

SECONDARY OUTCOMES:
Fail index | 48 months
  This outcome will be assessed by monitoring if the patient randomized did not fill the discharge criteria and/or needed a re-hospitalization
  There is no scale for this outcome; It will be reported by the percentage of patients that should be discharged in a specific day, but it was not discharged due to not fulfill one of the discharge criteria (adequate control of postoperative pain, absence of nausea and / or vomiting, absence of bleeding from the drain, being oriented, walking / walking without help from third parties and being able to ingest liquids properly, no hematúria, sero-urinary drainage rate up to 200 ml, no bleeding in the operative wound, release of light diet (liquid) after high anesthetic and recommendation of pasty diet (soups and liquids), prescription and standardization of analgesics and anti-inflammatory drugs (not on a demand schedule).
Factors that influence the patients' satisfaction: SATIS-BR | 48 months
  These outcomes will be evaluated through SATIS-BR questionnaire
  The unabbreviated scale name is "Escala da avaliação da satisfação dos usuários " ("Scale of evaluation of satisfaction of patients", in free English). The questionnaire contains 39 questions, with possible answers arranged in a Likert scale of 5 points, in which the value 1 indicates the lowest degree of satisfaction (worst outcome) and the value 5 indicates the highest degree of satisfaction (best outcome) with the service. The analysis will be performed in each question individually. The comparison of each question among groups will be performed using Analysis of Variance (ANOVA). Subsequently, Linear Regression will be used to verify the joint relationship among the characteristics of patients with the group influencing satisfaction.
  Additionally, there are 5 qualitative questions that will be analyzed in relation to factors that influence hospital stay and factors that influence the patients' satisfaction.
Assessment of how the patient feels about early discharge through an inventory | 48 months
  The inventory was created by the autors in order to evaluate patient´s satisfaction and perception of security, using the specific questions (here, translated to English):
  * What do you think about the hospitalization time in relation to the surgery?
  * Would you like to have been hospitalized any longer?
  * Are you satisfied with the type of anesthesia used in your surgery?
  * After the surgery, how did you feel about the medication prescribed for pain?
  * Did you feel satisfied with the explanation of the hospital discharge?
  * In general, how did you feel about satisfaction? The scale has answers arranged in a Likert scale of 5 points, in which the value 1 indicates the lowest degree of satisfaction (worst outcome) and the value 5 indicates the highest degree of satisfaction (best outcome). Each question will be analyzed individually. The perception of safety will be compared among the groups using the Chi-Square test (or Fisher's Exact).
Questionnaire assessing the patient´s satisfaction levels regarding the length of hospital stay | 48 months
  This outcome will be evaluated through SATIS-BR questionnaire
  The unabbreviated scale name is "Escala da avaliação da satisfação dos usuários " ("Scale of evaluation of satisfaction of patients", in free English). The questionnaire contains 39 questions, with possible answers arranged in a Likert scale of 5 points, in which the value 1 indicates the lowest degree of satisfaction (worst outcome) and the value 5 indicates the highest degree of satisfaction (best outcome) with the service. The analysis will be performed in each question individually. The comparison of each question among groups will be performed using Analysis of Variance (ANOVA). Subsequently, Linear Regression will be used to verify the joint relationship among the characteristics of patients with the group influencing satisfaction.
  Additionally, there are 5 qualitative questions that will be analyzed in relation to factors that influence hospital stay and factors that influence the patients' satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Eliney F Faria, MD, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Nucleo de Apoio ao Pesquisador, Barretos, São Paulo, Brazil

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT03674996/Prot_SAP_000.pdf